CLINICAL TRIAL: NCT02820116
Title: An Open-label, Multicenter，Single-arm, Phase II Clinical Study of Icotinib for IIIA - IIIB NSCLC Patients With Epidermal Growth Factor Receptor Mutation
Brief Title: The Role of Icotinib in the Perioperative Treatment of IIIA - IIIB NSCLC Patients With EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Haidian Hospital (Other)
Collaborators: Peking University People's Hospital (Other); 307 Hospital of PLA (Other); 309th Hospital of Chinese People's Liberation Army (Other)
Responsible Party: Principal Investigator, Huang Yuqing, Deputy Director, Beijing Haidian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIPOT1606
Record Dates: First submitted 2016-06-22; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer(NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib (Experimental): Patients receive Icotinib PO TID for 8 weeks and then undergo thoracotomy.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — In the neoadjuvant treatment phase, eligible patients will receive 125mg of Icotinib three times per day for 8 weeks (56 days). In the post-surgery phase, Icotinib 125mg/three tims/day taken orally for 2 years or till disease progression or unacceptable toxicity.
  Other Names: Conmana

SUMMARY:
This is an open-label, multicenter, single-arm, phase II interventional clinical trial evaluating efficacy and safety of Icotinib as neoadjuvant treatment in patients with IIIA- IIIB NSCLC with activating EGFR mutation in exon 19 or 21. Sixty-seven resectable stage IIIA- IIIB NSCLC patients with EGFR activating (19/21) mutations will be eligible to be enrolled. EGFR mutation will be prospectively tested in all the participants' biopsy samples and confirmed in surgical resected samples.

Neoadjuvant treatment phase:

Eligible patients will receive 125mg of Icotinib three times per day. Treatment will be scheduled to continue until the disease progression or unbearable toxicities appear.

Surgery treatment phase:

Tumor response will be evaluated with CT scan after 8 weeks of induction treatment. The patients with responsive disease considered to be technique resectable will undergo resection.

Post-surgery phase:

It is the discretion of the investigator whether the patient is a candidate for post-operative treatment which is considered to be in the best interest of the patients. It is recommended that patients with positive margins or residual tumor after surgery should receive radiation therapy. Patients after surgery will receive long-term follow-up -- chest CT scan，abdominal abdominal ultrasound every 3 months, brain MRI every 6 months, bone scan (ECT) every 12 months -- for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Pathologically confirmed non-small cell lung cancer with EGFR exon 19 deletion or exon 21 L858 mutation.
3. Clinically or pathologically confirmed stage IIIA- IIIB
4. Tolerable to complete resection of lung cancer
5. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications
6. ECOG performance status 0-1.
7. Life expectancy ≥12 weeks.
8. Measurable disease must be characterized according to RECIST 1.1 criteria. Measurable lesions are defined as those that can be accurately measured in at least one dimension as ≥ 10mm by spiral CT scan.
9. Adequate hematological function: Absolute neutrophil count (ANC) ≥2.0 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥10 g/dL (may be transfused to maintain or exceed this level).
10. Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN); Aspartate amino transferase (AST) and alanine amino transferase (ALT) ≤ 2.5 x upper limit of normal (ULN).
11. Adequate renal function: Serum creatinine ≤ 1.25 x upper limit of normal (ULN), and creatinine clearance≥ 60 ml/min.
12. Measurable disease according to the preset criteria .

Exclusion Criteria:

1. Patients with prior exposure to chemotherapy, irradiation or systemic anti-cancer therapy (e.g. monoclonal antibody therapy) for lung cancer.
2. Known severe hypersensitivity to Icotinib or any of the excipients of this product
3. Previous or current malignancies of other histologies within the last 5 years with the exception of the following: other malignancies cured by surgery alone and having a continuous disease-free survival of 5 years; cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix.
4. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within six months, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
5. Interstitial lung disease(ILD) or pulmonary fibrosis; impaired pulmonary function.
6. Eye inflammation or eye infection not fully treated or predisposing factor of this.
7. Uncontrolled central nervous system (CNS) metastasis.
8. Any serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study
9. Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the subject at high risk for treatment-related complications.
10. Pregnancy or breast feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2016-05; Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Complete resection rate | Complete resection rate is depended on the pathology diagnosis after surgery, an expected average of 8 weeks from enrollment.

SECONDARY OUTCOMES:
Objective response rate(ORR, i.e., complete response [CR] + partial response [PR]) | Up to 5 years
Disease control rate (CR + PR+ stable disease) | Up to 5 years
Clinical down-staging | 8 weeks
Progression free survival (PFS) | Participants after surgery will receive long-term follow-up for up to 5 years
Overall survival (OS) | Participants after surgery will receive long-term follow-up for up to 5 years
Number of Adverse Event | Within 28 days of last study dose

CONTACTS AND LOCATIONS:
Overall Officials: Jun liu, doctor, Principal Investigator — Peking University People Hospital
Locations (1):
- Beijing Haidian Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided